CLINICAL TRIAL: NCT00047697
Title: Donepezil HCl: Treating Cognitive Deficits in Autism
Brief Title: Donepezil HCl & Cognitive Deficits in Autism
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Benjamin L Handen, PhD, BCBA-D, Assistant Professor of Psychiatry & Pediatric, University of Pittsburgh
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R21MH064941 (NIH); R21MH064941 (NIH); DSIR CT-M3 (Other: NIMH)
Record Dates: First submitted 2002-10-11; First posted 2002-10-16 (Estimated); Results first posted 2017-10-05 (Actual); Last update posted 2017-10-05 (Actual); Status verified 2017-09

CONDITIONS: Autistic Disorder
MeSH Terms: conditions — Autistic Disorder | interventions — Donepezil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Donepezil HCl (Experimental): Donepezil HCL 5 mg and 10 mg
  Interventions: Drug: Donepezil HCl
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Donepezil HCl — Participants will start with 5 mg per day dose of donepezil HCl, then have their dose increased to 10mg per day after 4 weeks.
  Other Names: Aricept
  Arms: Donepezil HCl
Drug: Placebo — Placebo used in placed of Donepezil HCL
  Arms: Placebo

SUMMARY:
This 11-week study will examine the safety and effectiveness of the medication donepezil (Aricept®) compared to placebo for treating cognitive deficits in children and adolescents with Autism Spectrum Disorder.

DETAILED DESCRIPTION:
Children with autism spectrum disorder (ASD) often have impaired communication, problems with social interaction, and repetitive and stereotyped patterns of behavior. While most research has attempted to treat the behavioral deficits commonly associated with ASD, few studies have attempted to improve the core features of this disorder. A recent study found that donepezil HCl helped to improve speech production, attention span, and ability to express emotions in a group of children with autism. This study will provide an opportunity to conduct further testing of the effects of donepezil HCl on the cognitive deficits presumed to underlie the core features of ASD.

This study begins at Week 1 with a baseline assessment. Participants are then randomly assigned to either donepezil HCl or placebo. Participants will start with either a 5mg/day dose of donepezil HCl or placebo followed by a cognitive assessment after 4 weeks on this dose. Participants will then have their dose increased to 10mg/day. Another cognitive assessment will be given after 4 weeks on this dose.

ELIGIBILITY:
Inclusion Criteria:

* Autism Spectrum Disorder (ASD)
* Asperger's Disorder
* IQ of 75 or above
* Baseline assessment tests within the acceptable range

Exclusion Criteria:

* Bipolar disorder, schizophrenia, schizoaffective disorder, or psychotic disorder
* Seizure disorder requiring the use of anticonvulsant medications
* Congenital rubella, cytomegalovirus, or tuberous sclerosis
* Certain medications prescribed for management of behavior (please contact the investigator for a complete list)
* Medications/preparations that are known to interact with donepezil HCl
* Significant medical illness, endocrinopathies, cardiovascular disease, or severe chronic malnutrition
* Pregnancy or sexually active females not using a reliable method of contraception

Ages: 8 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2002-10; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin L. Handen, PhD, Principal Investigator — University of Pittsburgh, School of Medicine, Department of Psychiatry
Locations (1):
- Western Psychiatric Institute & Clinic, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No
We have no specific plan to share data at this time.

RESULTS

PARTICIPANT FLOW:
Groups:
- Donepezil HCL: Subjects placed on 5 and 10 mg of donepezil
- Placebo: Subjects placed on 5 mg or 10 mg of placebo
Period: Overall Study
Arm/Group | Donepezil HCL | Placebo
Started | 18 | 16
Completed | 18 | 14
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Participants will start with 5 mg/day of placebo, then have their doses increased to 10 mg/day of placebo after 4 weeks.
- Total: Total of all reporting groups
Arm/Group | Donepezil HCL | Placebo | Total
Number analyzed (Participants) | 18 | 16 | 34
Age, Continuous [Mean (Full Range); unit: years] | 11.6 [8.7 to 16.8] | 11.8 [8.1 to 16.6] | 11.7 [8.1 to 16.8]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 17 | 14 | 31
Cognitive Assessment: TMT [Mean (Standard Deviation); unit: Seconds] — TMT: Trial-Making Test. Time (sec) Range: 0 - 300. Lower = better
  Seconds | 123.6 (56.5) | 154.9 (77.8) | 138.3 (66.5)
Cognitive Assessment: EOWVT Standard score [Mean (Standard Deviation); unit: units on a scale] — Expressive One Word Vocabulary Test (standard score) Range: 55-140. Higher = better
  units on a scale | 104.6 (22.4) | 108.7 (17.0) | 106.5 (19.9)
Cognitive Assessment: CVLT [Mean (Standard Deviation); unit: Correct answers, percentage] — California Verbal Learning Test (percent of correct answers) Range: 0-100. Higher = better
  Correct answers, percentage | 40.7 (14.1) | 47.1 (10.3) | 43.7 (12.3)

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Assessment: TMT
Description: TMT: Trial-Making Test. Time (sec) Range: 0 - 300. Lower = better
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Donepezil HCl | Placebo
Number analyzed (Participants) | 18 | 16
seconds | 118.3 (79.1) | 104.7 (53.4)

2. Primary Outcome: Cognitive Assessment: EOWVT Standard Score
Description: Expressive One Word Vocabulary Test (standard score) Range: 55-140. Higher = better
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Placebo used in place of Donepezil HCL
Arm/Group | Donepezil HCl | Placebo
Number analyzed (Participants) | 18 | 16
units on a scale | 109.7 (21.0) | 114.5 (16.1)

3. Primary Outcome: Cognitive Assessment: CVLT
Description: California Verbal Learning Test (percent of correct answers) Range: 0-100. Higher = better
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: percentage of correct answers
Arm/Group | Donepezil HCl | Placebo
Number analyzed (Participants) | 18 | 16
percentage of correct answers | 50.2 (11.0) | 51.3 (14.7)

ADVERSE EVENTS:
Time Frame: AEs were collected for 10 weeks (and for longer if a subject had an active AE at the end of the 10-week trial).
Groups:
- Donepezil HCL: 5 mg of donepezil for 4 weeks, followed by 10 mg of donepezil for 6 weeks.
- Placebo: Placebo substituted for Donepezil HCL
Arm/Group | Donepezil HCL | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 0/18 | 0/16

LIMITATIONS AND CAVEATS:
The trial may not have been long enough to obtain clinically significant effects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No